CLINICAL TRIAL: NCT06429969
Title: Nuclear Magnetic Resonance (NMR)-Based Metabolomic Characterisation of Vitreoretinal Diseases Using Vitreous Fluid
Brief Title: Metabolomic Profile of Vitreoretinal Diseases: an NMR-Based Approach Using Vitreous.
Acronym: NMR
Status: Recruiting | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: WDRY2022-K222
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-01

CONDITIONS: Vitreoretinal Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The vitreous body is a transparent gel composed mainly of fibrous collagen and hydrophilic hyaluronic acid, with a volume of approximately 4.5 ml, constituting the largest volume in the eye. When patients suffer from vitreoretinal diseases such as IMH, DR, RD, IMM, RVO, PPV is usually required so that it can constitute a passageway to allow instruments to enter the retina for manipulation, at which point the vitreous is disposed of as waste.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- IMH group: Participants diagnosed with idiopathic macular hole(IMH) requiring PPV were enrolled in the IMH group, and this group was a control group because the vitreous of IMH may be closest to normal and normal people do not undergo PPV. 100-250ul of vitreous fluid was collected intraoperatively for NMR analysis.
- DR group: In patients with a confirmed diagnosis of diabetic retinopathy (DR) and requiring PPV surgery, 100-250ul of vitreous fluid was collected intraoperatively for NMR analysis.
- RD group: In patients with a confirmed diagnosis of retinal detachment (RD) and requiring PPV surgery, 100-250ul of vitreous fluid was collected intraoperatively for NMR analysis.
- IMM group: In patients with a confirmed diagnosis of idiopathic macular epiretinal membrane (IMM) and requiring PPV surgery, 100-250ul of vitreous fluid was collected intraoperatively for NMR analysis.
- RVO group: In patients with a confirmed diagnosis of retinal vein occlusion (RVO) and requiring PPV surgery, 100-250ul of vitreous fluid was collected intraoperatively for NMR analysis.

SUMMARY:
The goal of this observational study was to learn about metabolomics profiles in vitreoretinal diseases by nuclear magnetic resonance (NMR)using vitreous fluid. The main question it aimed to answer was abnormal biomarkers for common retinal diseases such as idiopathic macular hole(IMH), diabetic retinopathy(DR) and retinal detachment(RD). Participants would not be subjected to any intervention and the investigators would only collect preoperative information and remaining vitreous samples. The investigators divided the participants into groups with appropriate disease names based on the disease diagnosis, such as IMH group, DR group, and RD group. The MH group was used as a control group, investigators compared other groups to see the metabolomic abnormalities.

DETAILED DESCRIPTION:
This study aimed to analyze vitreous fluid using NMR to discover potential biomarkers for the prevention, early diagnosis, and treatment of vitreoretinal diseases and to reveal the mechanisms of disease progression. Patients suffering from IMH, DR, RD, idiopathic macular epiretinal membrane (IMM), and retinal vein occlusion (RVO) quiring for pars plana vitrectomy (PPV), who visited Renmin Hospital of Wuhan University, were chosen to participate in this study. Participants were not subjected to any intervention and the investigator only collected preoperative information and remaining vitreous samples. Participants provided preoperative examination information and medical history, and the investigators divided the participants into five groups with corresponding disease names based on the disease diagnosis, including five groups for five diseases: IMH group, DR group, RD group, IMM group, and RVO group. The control group for the diseases was the IMH group, and metabolomic differences were observed. These patients are usually treated with PPV, during PPV typically performed on these patients, vitreous fluid is usually disposed of as waste, and investigators collected 100-250 ul of the fluid for NMR analysis to see metabolomic characterization of these diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of IMH diagnosis with concomitant need for PPV surgery;
2. Confirmation of DR diagnosis with concomitant need for PPV surgery;
3. Confirmation of RD diagnosis with concomitant need for PPV surgery;
4. Confirmation of IMM diagnosis with concomitant need for PPV surgery;
5. Confirmation of RVO diagnosis with concomitant need for PPV surgery.

Exclusion Criteria:

1. Diagnosed vitreoretinal disease with no need for PPV surgery;
2. Previous history of PPV surgery;
3. Combination of other active ophthalmic diseases, such as acute conjunctivitis and uveitis;
4. Combination of serious systemic diseases such as hypertension and diabetes mellitus.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrolled participants were patients who attended Renmin Hospital of Wuhan University with a confirmed diagnosis of vitreoretinal disease. As a result, most of the participants were residents of Hubei Province, China. It is expected that vitreous fluid samples collected from patients with IMH, DR, RD, IMM, and RVO were 50, 100, 100, 50, and 50, respectively, for a total of 450, with about a mean age of 56 years.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2027-04-17 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative amino acid concentration(Unite: %) | intraoperative
  NMR provides spectral data to show the relative concentration of various amino acids, and the use of NMR to measure vitreous humor and compare changes in amino acid content across disease species leads to speculation about biological markers of disease progression.

SECONDARY OUTCOMES:
Relative concentrations of macromolecules such as glucose and lipids(Unite: %) | intraoperative
  Macromolecules such as glucose and lipids also play a role in the metabolism of vitreoretinal diseases, so NMR spectroscopy will be used to show the relative concentration of macromolecules.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Du, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Eye, Center, Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
This is not considered for the time being, as further processing of the samples are required subsequently and there may be culling data.